CLINICAL TRIAL: NCT01364883
Title: A Phase I Study to Assess the Safety and Immunogenicity of Novel Schedules for Vaccination With the Candidate Malaria Vaccines AdCh63 ME-TRAP and MVA ME-TRAP
Brief Title: Safety and Immunogenicity of Novel Vaccination Schedules With Malaria Vaccines AdCh63 ME-TRAP and MVA ME-TRAP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAC043
Record Dates: First submitted 2011-05-31; First posted 2011-06-03 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: Malaria
Keywords: Vaccine; Immune response
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Group 1 (Experimental): AdCh63 ME-TRAP prime D0, AdCh63 ME-TRAP boost W4, AdCh63 ME-TRAP boost W8, MVA ME-TRAP boost W16
  Interventions: Biological: Vaccination Schedule One
- Group 2 (Experimental): AdCh63 ME-TRAP prime D0, AdCh63 ME-TRAP boost W8, MVA ME-TRAP boost W16, MVA ME-TRAP boost W24
  Interventions: Biological: Vaccination Schedule Two
- Group 3 (Experimental): AdCh63 ME-TRAP prime D0, AdCh63 ME-TRAP boost W4, MVA ME-TRAP boost W8, MVA ME-TRAP boost W12
  Interventions: Biological: Vaccination Schedule Three
- Group 4 (Experimental): AdCh63 ME-TRAP prime D0, MVA ME-TRAP boost W8, MVA ME-TRAP boost W16, MVA ME-TRAP boost W24
  Interventions: Biological: Vaccination Schedule Four
- Group 5 (Experimental): AdCh63 ME-TRAP prime D0, MVA ME-TRAP boost W4, AdCh63 ME-TRAP boost W8, MVA ME-TRAP boost W16
  Interventions: Biological: Vaccination Schedule Five
- Group 6 (Experimental): AdCh63 ME-TRAP prime D0, MVA ME-TRAP boost W4, AdCh63 ME-TRAP boost W8, MVA ME-TRAP boost W12
  Interventions: Biological: Vaccination Schedule Six
- Group 7 (Experimental): AdCh63 ME-TRAP prime D0, MVA ME-TRAP boost W8, AdCh63 ME-TRAP boost W16, MVA ME-TRAP boost W24
  Interventions: Biological: Vaccination Schedule Seven

INTERVENTIONS:
Biological: Vaccination Schedule One — Intramuscular injection of 5x10^10 vp of AdCh63 ME-TRAP, intramuscular injection of 2x10^8 pfu of MVA ME-TRAP
  Arms: Group 1
Biological: Vaccination Schedule Two — Intramuscular injection of 5x10^10 vp of AdCh63 ME-TRAP, intramuscular injection of 2x10^8 pfu of MVA ME-TRAP
  Arms: Group 2
Biological: Vaccination Schedule Three — Intramuscular injection of 5x10^10 vp of AdCh63 ME-TRAP, intramuscular injection of 2x10^8 pfu of MVA ME-TRAP
  Arms: Group 3
Biological: Vaccination Schedule Four — Intramuscular injection of 5x10^10 vp of AdCh63 ME-TRAP, intramuscular injection of 2x10^8 pfu of MVA ME-TRAP
  Arms: Group 4
Biological: Vaccination Schedule Five — Intramuscular injection of 5x10^10 vp of AdCh63 ME-TRAP, intramuscular injection of 2x10^8 pfu of MVA ME-TRAP
  Arms: Group 5
Biological: Vaccination Schedule Six — Intramuscular injection of 5x10^10 vp of AdCh63 ME-TRAP, intramuscular injection of 2x10^8 pfu of MVA ME-TRAP
  Arms: Group 6
Biological: Vaccination Schedule Seven — AdCh63 ME-TRAP prime D0, AdCh63 ME-TRAP boost W8, AdCh63 ME-TRAP boost W16, MVA ME-TRAP boost W24
  Arms: Group 7

SUMMARY:
This is an open label phase I study, to assess the safety and immunogenicity of novel schedules for vaccination with the candidate malaria vaccines AdCh63 ME-TRAP and MVA ME-TRAP. These vaccines have been evaluated previously in a number of clinical trials proved to be safe and capable of inducing protective cellular immune response following challenge with the parasite. All volunteers recruited will be healthy adults. They will be primed with AdCh63 ME-TRAP administered intramuscularly and boosted several times with AdCh63 ME-TRAP and MVA ME-TRAP according to various schedules.. Safety data will be collected for each of the seven regimens. Secondary aims of this study will be to assess the immune responses generated by each of these regimes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 50 years
* Able and willing (in the Investigator's opinion) to comply with all study requirements
* Willing to allow the investigators to discuss their medical history with their General Practitioner
* For female volunteers, willingness to practice continuous effective contraception during the study
* Agreement to refrain from blood donation during the course of the study
* Written informed consent

Exclusion Criteria:

* Participation in another research study involving an investigational product in the 30 days preceding enrolment, or planned use during the study period
* Prior receipt of an investigational malaria vaccine or any other investigational vaccine likely to impact on interpretation of the trial data
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
* Pregnancy, lactation, or intention to become pregnant during the study
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, e.g. egg products, Kathon History of clinically significant contact dermatitis
* Any history of anaphylaxis in relation to vaccination
* Any history of malaria Travel to a malaria endemic region during the study period or within the six months preceding enrolment in the study
* History of serious psychiatric condition that may affect participation in the study
* Any other serious chronic illness requiring hospital specialist supervision -Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
* Suspected or known injecting drug abuse in the five years preceding enrolment -Seropositive for hepatitis B surface antigen (HBsAg)
* Seropositive for hepatitis C virus (antibodies to HCV)
* Any relevant history of cancer (excludes basal cell carcinoma of the skin and cervical carcinoma in situ)
* Any clinically significant abnormal finding on screening biochemistry or haematology blood tests or urinalysis
* Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of study data

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2011-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Vaccine Safety | Participants will be followed for the duration of the study, an expected average of 21 months
  To assess the safety of vaccination of healthy adults with AdCh63 ME-TRAP and MVA ME-TRAP according to vaccination schedules 1 to 7

SECONDARY OUTCOMES:
Vaccine immunogenicity | Participants will be followed for the duration of the study, an expected average of 21months
  To assess the immunogenicity of vaccination of healthy adults with AdCh63 ME-TRAP and MVA ME-TRAP according to vaccination schedules 1 to 7

CONTACTS AND LOCATIONS:
Overall Officials: Adrian VS Hill, Principal Investigator — University of Oxford
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, University of Oxford, Oxford, United Kingdom